CLINICAL TRIAL: NCT02974621
Title: A Randomized Phase 2 Trial of Cediranib and Olaparib Compared to Bevacizumab in Patients With Recurrent Glioblastoma Who Have Not Received Prior VEGF Therapy
Brief Title: Cediranib Maleate and Olaparib Compared to Bevacizumab in Treating Patients With Recurrent Glioblastoma
Status: Active, not recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: NCI-2016-01769; NCI-2016-01769 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); 17-735; 10067 (Other: Dana-Farber - Harvard Cancer Center LAO); 10067 (Other: CTEP); UM1CA186709 (NIH)
Record Dates: First submitted 2016-11-23; First posted 2016-11-28 (Estimated); Results first posted 2024-02-02 (Actual); Last update posted 2025-08-03 (Actual); Status verified 2025-07

CONDITIONS: Recurrent Glioblastoma
MeSH Terms: conditions — Glioblastoma | interventions — Bevacizumab; Immunoglobulin G; Disulfides; cediranib; olaparib

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Arm A (olaparib, cediranib maleate) (Experimental): Patients receive olaparib PO BID and cediranib maleate PO once QD on days 1-28. Cycles repeat every 28 days in the absence of disease progression or unacceptable toxicity.
  Interventions: Drug: Cediranib; Drug: Cediranib Maleate; Drug: Olaparib
- Arm B (bevacizumab) (Experimental): Patients receive bevacizumab IV over 30-90 minutes every 2 weeks. Cycles repeat every 28 days in the absence of disease progression or unacceptable toxicity.
  Interventions: Biological: Bevacizumab

INTERVENTIONS:
Biological: Bevacizumab — Given IV
  Other Names: ABP 215; ABP-215; ABP215; Alymsys; Anti-VEGF; Anti-VEGF Humanized Monoclonal Antibody; Anti-VEGF Monoclonal Antibody SIBP04; Anti-VEGF rhuMAb; Avastin; Avzivi; Aybintio; BAT 1706; BAT-1706; BAT1706; BAT1706 Biosimilar; Bevacizumab awwb; Bevacizumab Biosimilar ABP 215; Bevacizumab Biosimilar BAT1706; Bevacizumab Biosimilar BEVZ92; Bevacizumab Biosimilar BI 695502; Bevacizumab Biosimilar CBT 124; Bevacizumab Biosimilar CT-P16; Bevacizumab Biosimilar FKB238; Bevacizumab Biosimilar GB-222; Bevacizumab Biosimilar HD204; Bevacizumab Biosimilar HLX04; Bevacizumab Biosimilar IBI305; Bevacizumab Biosimilar LY01008; Bevacizumab Biosimilar MB02; Bevacizumab Biosimilar MIL60; Bevacizumab Biosimilar Mvasi; Bevacizumab Biosimilar MYL-1402O; Bevacizumab Biosimilar QL 1101; Bevacizumab Biosimilar QL1101; Bevacizumab Biosimilar RPH-001; Bevacizumab Biosimilar SCT501; Bevacizumab Biosimilar Zirabev; Bevacizumab-adcd; Bevacizumab-awwb; Bevacizumab-aybi; Bevacizumab-bvzr; Bevacizumab-equi; Bevacizumab-maly; Bevacizumab-onbe; Bevacizumab-tnjn; BP102; BP102 Biosimilar; CT P16; CT-P16; CTP16; Equidacent; FKB 238; FKB-238; FKB238; HD204; Immunoglobulin G1 (Human-Mouse Monoclonal rhuMab-VEGF Gamma-Chain Anti-Human Vascular Endothelial Growth Factor), Disulfide With Human-Mouse Monoclonal rhuMab-VEGF Light Chain, Dimer; MB 02; MB-02; MB02; Mvasi; MYL-1402O; Onbevzi; Oyavas; PF 06439535; PF-06439535; PF06439535; QL1101; Recombinant Humanized Anti-VEGF Monoclonal Antibody; rhuMab-VEGF; SCT501; SIBP 04; SIBP-04; SIBP04; Vegzelma; Zirabev
  Arms: Arm B (bevacizumab)
Drug: Cediranib — Given PO
  Other Names: AZ-D2171; AZD 2171; AZD2171
  Arms: Arm A (olaparib, cediranib maleate)
Drug: Cediranib Maleate — Given PO
  Other Names: AZD2171; AZD2171 Maleate; Recentin
  Arms: Arm A (olaparib, cediranib maleate)
Drug: Olaparib — Given PO
  Other Names: AZD 2281; AZD-2281; AZD2281; KU 0059436; KU-0059436; KU0059436; Lynparza; Olanib; Olaparix; PARP Inhibitor AZD2281
  Arms: Arm A (olaparib, cediranib maleate)

SUMMARY:
This randomized phase II trial studies how well cediranib maleate and olaparib work compared to bevacizumab in treating patients with glioblastoma that has come back (recurrent). Cediranib maleate and olaparib may stop the growth of tumor cells by blocking some of the enzymes needed for cell growth. Immunotherapy with monoclonal antibodies, such as bevacizumab, may help the body's immune system attack the cancer, and may interfere with the ability of tumor cells to grow and spread.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVES:

I. To compare the antitumor activity of cediranib maleate (cediranib)/olaparib versus reference bevacizumab monotherapy, as measured by progression-free survival at 6 months (PF6), in patients with recurrent glioblastoma (GBM).

SECONDARY OBJECTIVES:

I. To compare overall survival (OS), progression free survival (PFS) and objective response (ORR) in patients with recurrent GBM treated with cediranib/olaparib versus bevacizumab.

II. To assess the safety of the combination of olaparib and cediranib in patients with recurrent GBM.

III. To evaluate the association of blood based biomarkers involved with angiogenesis using the Biomarker Review Committee-approved Plasma Angiome Panel (bFGF, Ang-1, Ang-2, Tie-2, SDF1-alpha, Collagen IV, PlGF, sVEGFR1, sVEGFR2, VEGF, Il-1beta, Il-6, Il-8, TNF-alpha, CAIX) with the clinical activity of cediranib/olaparib.

IV. To evaluate the association of tissue biomarkers involved with deoxyribonucleic acid (DNA) repair using the Biomarker Review Committee-approved BROCA panel with the clinical activity of cediranib/olaparib.

V. To identify genomic alteration by whole exome sequencing in GBM tumor specimens that correlate with the clinical activity of cediranib/olaparib.

VI. To evaluate the association of magnetic resonance imaging (MRI) imaging parameters (tumor perfusion and oxygenation, brain tumor cellularity) with the biological response of cediranib/olaparib.

VII. To contribute genetic analysis data from de-identified biospecimens to Genomic Data Commons (GDC), a well annotated cancer molecular and clinical data repository, for current and future research; specimens will be annotated with key clinical data, including presentation, diagnosis, staging, summary treatment, and if possible, outcome.

VIII. To bank formalin-fixed, paraffin-embedded (FFPE) tissue, blood (for cell-free DNA analysis), and nucleic acids obtained from patients at the Experimental Therapeutics Clinical Trials Network (ETCTN) Biorepository at Nationwide Children's Hospital.

OUTLINE: Patients are randomized to 1 of 2 arms.

ARM A: Patients receive olaparib orally (PO) twice daily (BID) and cediranib maleate PO once daily (QD) on days 1-28.

ARM B: Patients receive bevacizumab intravenously (IV) over 30-90 minutes every 2 weeks.

In both arms, cycles repeat every 28 days in the absence of disease progression or unacceptable toxicity.

After completion of study treatment, patients are followed up at 30 days and then periodically for 3 years.

ELIGIBILITY:
Inclusion Criteria:

* Unequivocal evidence of progressive disease on contrast-enhanced brain computed tomography (CT) or MRI as defined by Response Assessment in Neuro-Oncology (RANO) criteria, or have documented recurrent glioblastoma on diagnostic biopsy
* Previous therapy with at least radiotherapy and temozolomide
* Must be 12 weeks from radiotherapy; if patients are within 12 weeks of radiotherapy, then the progressive lesion must be outside of the high-dose radiation target volume or have unequivocal evidence of progressive tumor on a biopsy specimen
* Only first and second recurrences of GBM are eligible
* From the projected start of scheduled study treatment, the following time periods must have elapsed: 5 half-lives from investigational agents, 4 weeks from cytotoxic therapy (except 23 days for temozolomide and 6 weeks from nitrosoureas), 6 weeks from antibodies, or 4 weeks (or 5 half-lives, whichever is shorter) from other systemic anti-tumor therapies; treatment on study may start one day after discontinuation of the optune device
* All adverse events grade > 1 related to prior therapies (chemotherapy, radiotherapy, and/or surgery) must be resolved, except for alopecia
* Willingness to release archival tissue sample for research purposes, if available
* Karnofsky performance status >= 60
* Life expectancy of at least 3 months
* Leukocytes >= 3,000/mcL
* Absolute neutrophil count >= 1,500/mcL
* Platelets >= 100,000/mcL
* Hemoglobin >= 10.0 g/dL and no blood transfusions in the 28 days prior to entry/randomization
* Total bilirubin =< 1.5 x institutional upper limit of normal (ULN)
* Aspartate aminotransferase (AST) (serum glutamic-oxaloacetic transaminase [SGOT])/alanine aminotransferase (ALT) (serum glutamate pyruvate transaminase [SGPT]) =< 2.5 x institutional upper limit of normal
* Creatinine should not exceed the institutional upper limit of normal OR creatinine clearance >= 60 mL/min/1.73 m^2
* Urine protein: creatinine (UPC) ratio < 1 or urine dipstick for proteinuria =< 2+ (note: if the UPC ratio is >= 1.0 then a 24-hour urine collection should be performed and this must demonstrate =< 1 g of protein in 24 hours)
* CT or MRI within 14 days prior to start of study drug
* Corticosteroid dose must be stable or decreasing for at least 5 days prior to the baseline MRI scan
* The effects of olaparib and cediranib on the developing human fetus are unknown; female subjects must either be of non-reproductive potential, not breast-feeding or must have a negative urine or serum pregnancy test within 28 days of study treatment, confirmed prior to treatment on day 1; women of child-bearing potential and men must agree to use adequate contraception (hormonal or barrier method of birth control; abstinence) prior to study entry and for the duration of study participation; should a woman become pregnant or suspect she is pregnant while she or her partner is participating in this study, she should inform her treating physician immediately; men treated or enrolled on this protocol must also agree to use adequate contraception prior to the study, for the duration of study participation, and 6 months after completion of olaparib + cediranib administration
* Ability to understand and the willingness to sign a written informed consent document

Exclusion Criteria:

* Participants should not have received any other investigational agents nor have participated in an investigational trial within the past 4 weeks
* Participants may not have had prior use of PARP inhibitors; patients may not have received prior treatment affecting the VEGF pathway including but not limited to thalidomide, bevacizumab, sunitinib, or sorafenib
* Patients who are receiving any other investigational agents
* History of allergic reactions attributed to compounds of similar chemical or biologic composition to olaparib, cediranib or bevacizumab
* Participants may not have any evidence of ongoing inadequately controlled hypertension (defined as a systolic blood pressure [BP] of > 140 mmHg or a diastolic BP of > 90 mmHg); patients with hypertension may not be on more than three antihypertensive medications for management of their blood pressure (medications that combine two anti-hypertensives into one are considered as two medications); it is strongly recommended that patients who require three antihypertensive medications for baseline management of pre-existing hypertension be actively followed by a cardiologist or blood pressure specialist for management of BP while on protocol
* Participants may not have had any prior history of hypertensive crisis or hypertensive encephalopathy
* Participants may not have had history of abdominal fistula or gastrointestinal perforation within the past 6 months
* Participants may not have had a history of intra-abdominal abscess within the past 6 months
* Patients may not have a known or confirmed history of pneumonitis
* Participants may not have current signs and/or symptoms of bowel obstruction or signs and/or symptoms of bowel obstruction within 3 months prior to starting study drugs
* Participants may not have a dependency on IV hydration or total parenteral nutrition (TPN)
* Patients with myelodysplastic syndrome/acute myeloid leukemia
* Participants with any concomitant or prior invasive malignancies are ineligible with the following exceptions:

  * Treated limited-stage basal cell or squamous cell carcinoma of the skin
  * Carcinoma in situ of the breast or cervix
  * Prior cancer treated with curative intent with no evidence of recurrent disease 3 years following diagnosis and judged by the investigator to be at low risk of recurrence
* Participants with any of the following:

  * History of myocardial infarction within six months
  * Unstable angina
  * History of cerebrovascular accident (CVA) within 6 months
  * New York Heart Association grade II or greater congestive heart failure
  * Significant vascular disease (e.g. aortic aneurysm, history of aortic dissection)
  * Clinically significant peripheral vascular disease
* If cardiac function assessment is clinically indicated or performed: participants will be ineligible if left ventricular ejection fraction (LVEF) is less than normal per institutional guidelines, or < 55%, if the threshold for normal is not otherwise specified by institutional guidelines
* Participants may not have corrected QT (QTc) > 470 msec or family history of long QT syndrome
* Participants may not have a major surgical procedure, open biopsy, or significant traumatic injury within 28 days prior to starting cediranib; anticipation of need for major surgical procedures during the course of the study also excludes patients from the trial
* Participants should not have any uncontrolled intercurrent illness including, but limited to ongoing or active infection, symptomatic congestive heart failure, unstable angina pectoris, cardiac arrhythmia, or psychiatric illness/social situations that would limit compliance with study requirements
* Participants receiving any medications or substances that are strong inhibitors or inducers of CYP3A4 or moderate inhibitors of CYP3A4 are ineligible; the study team should check a frequently-updated medical reference for a list of drugs to avoid or minimize use of; as part of the enrollment/informed consent procedures, the patient will be counseled on the risk of interactions with other agents, and what to do if new medications need to be prescribed or if the patient is considering a new over-the-counter medicine or herbal product; dihydropyridine calcium-channel blockers are permitted for management of hypertension; patient drug information handout and wallet card should be provided to patients
* Pregnant women are excluded from this study because cediranib and olaparib agent with the potential for teratogenic or abortifacient effects; because there is an unknown but potential risk for adverse events in nursing infants secondary to treatment of the mother with cediranib and olaparib breastfeeding should be discontinued if the mother is treated with cediranib and olaparib; these potential risks may also apply to other agents used in this study
* Human immunodeficiency virus (HIV)-positive patients on combination antiretroviral therapy are ineligible because of the potential for pharmacokinetic interactions with cediranib and olaparib; in addition, these patients are at increased risk of lethal infections when treated with marrow-suppressive therapy; appropriate studies will be undertaken in patients receiving combination antiretroviral therapy when indicated
* Current use of a prohibited medication; the following medications or non-drug therapies are prohibited:

  * Other anti-cancer therapy while on study treatment
  * Concurrent treatment with bisphosphonates is permitted; however, treatment must be initiated prior to the first dose of study therapy; prophylactic use of bisphosphonates in patients without bone disease is not permitted, except for the treatment of osteoporosis
  * Because the composition, pharmacokinetics (PK), and metabolism of many herbal supplements are unknown; the concurrent use of all herbal supplements is prohibited during the study (including, but not limited to, cannabis, S. John's wort, kava, ephedra [ma huang], gingko biloba, dehydroepiandrosterone [DHEA], yohimbe, saw palmetto or ginseng)
  * Raloxifene is allowed for patients taking it for bone health
* Participants should not have evidence of coagulopathy or bleeding diathesis; therapeutic anticoagulation for prior thromboembolic events is permitted

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 70 (Actual)
Dates: Start 2017-12-07 (Actual); Primary Completion 2022-12-31 (Actual); Study Completion 2026-07-17 (Estimated)

CONTACTS AND LOCATIONS:
Overall Officials: Isabel Arrillaga-Romany, Principal Investigator — Dana-Farber - Harvard Cancer Center LAO
Locations (27):
- United States (27):
  - UC San Diego Moores Cancer Center, La Jolla, California
  - UCHealth University of Colorado Hospital, Aurora, Colorado
  - Smilow Cancer Hospital-Derby Care Center, Derby, Connecticut
  - Smilow Cancer Hospital Care Center-Fairfield, Fairfield, Connecticut
  - Smilow Cancer Hospital Care Center - Guilford, Guilford, Connecticut
  - Smilow Cancer Hospital Care Center at Saint Francis, Hartford, Connecticut
  - Smilow Cancer Center/Yale-New Haven Hospital, New Haven, Connecticut
  - Yale University, New Haven, Connecticut
  - Smilow Cancer Hospital-Orange Care Center, Orange, Connecticut
  - Smilow Cancer Hospital-Torrington Care Center, Torrington, Connecticut
  - Smilow Cancer Hospital Care Center-Trumbull, Trumbull, Connecticut
  - Smilow Cancer Hospital-Waterbury Care Center, Waterbury, Connecticut
  - Smilow Cancer Hospital Care Center - Waterford, Waterford, Connecticut
  - Moffitt Cancer Center, Tampa, Florida
  - University of Kentucky/Markey Cancer Center, Lexington, Kentucky
  - Massachusetts General Hospital Cancer Center, Boston, Massachusetts
  - Dana-Farber Cancer Institute, Boston, Massachusetts
  - Siteman Cancer Center at Saint Peters Hospital, City of Saint Peters, Missouri
  - Siteman Cancer Center at West County Hospital, Creve Coeur, Missouri
  - Washington University School of Medicine, St Louis, Missouri
  - Siteman Cancer Center-South County, St Louis, Missouri
  - Siteman Cancer Center at Christian Hospital, St Louis, Missouri
  - Rutgers Cancer Institute of New Jersey, New Brunswick, New Jersey
  - NYP/Columbia University Medical Center/Herbert Irving Comprehensive Cancer Center, New York, New York
  - Duke University Medical Center, Durham, North Carolina
  - Ohio State University Comprehensive Cancer Center, Columbus, Ohio
  - University of Pittsburgh Cancer Institute (UPCI), Pittsburgh, Pennsylvania

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Arm A (Olaparib, Cediranib Maleate) | Arm B (Bevacizumab)
Started | 35 | 35
Completed | 34 | 25
Not Completed | 1 | 10
Not completed — Didn't receive study treatment | 1 | 10

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Arm A (Olaparib, Cediranib Maleate) | Arm B (Bevacizumab) | Total
Number analyzed (Participants) | 35 | 35 | 70
Age, Continuous [Median (Full Range); unit: years] | 60.0 [27.0 to 77.0] | 61.0 [19.0 to 79.0] | 60.5 [19.0 to 79.0]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 14 | 13 | 27
  Male | 21 | 22 | 43
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 1 | 0 | 1
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 2 | 1 | 3
  White | 29 | 33 | 62
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 3 | 1 | 4
Karnofsky performance status [Count of Participants; unit: Participants] — Karnofsky performance scale (KPS) is an assessment tool for functional impairment. KPS scoring ranges from 0-100, where 0 means death and 100 means normal function with no complaints or evidence of disease. Participants are eligible for the study if they have KPS scores greater than or equal to 60. KPS score 60 means participants require occasional assistance, but are able to care for most of their needs.
  Participants
    Score = 100 | 3 | 6 | 9
    Score = 90 | 13 | 14 | 27
    Score = 80 | 12 | 7 | 19
    Score = 70 | 7 | 6 | 13
    Score = 60 | 0 | 2 | 2
Time from initial surgery to study randomization [Median (Full Range); unit: days] | 375 [29 to 3360] | 309 [123 to 1720] | 353 [29 to 3360]
Number of Disease Recurrence [Count of Participants; unit: Participants]
  1 recurrence | 22 | 27 | 49
  2 recurrences | 13 | 8 | 21
Surgery [Count of Participants; unit: Participants]
  Resection | 32 | 27 | 59
  Biopsy | 2 | 8 | 10
IDH mutation [Count of Participants; unit: Participants] — IDH mutation is a known prognostic molecular marker of glioblastoma.
  Participants
    Yes | 8 | 5 | 13
    No | 26 | 29 | 55
    Unknown | 1 | 1 | 2
MGMT promoter methylation [Count of Participants; unit: Participants] — MGMT promoter methylation is a known prognostic molecular marker of glioblastoma.
  Participants
    Methylated | 11 | 13 | 24
    Unmethylated | 15 | 12 | 27
    Indeterminate | 2 | 1 | 3
    Unknown | 7 | 9 | 16

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With Progression-Free Survival at 6 Months
Description: Progression-Free Survival (PFS) is defined as the time from randomization to progressive disease (PD) per Response Assessment in Neuro-Oncology (RANO) criteria, or death due to any cause, whichever occurs first. Participants alive without PD are censored at date of last disease evaluation.
  PD criteria:
  (A) 25% increase in sum of the products of perpendicular diameters of enhancing lesions (over best response or baseline if no decrease) on stable or increasing doses of steroids and/or one or more of the following: (B) Significant increase in T2/FLAIR non-enhancing lesion on stable or increasing doses of steroids compared to baseline scan or best response following initiation of therapy, not due to co-morbid events (C) Any new lesions (D) Clear clinical deterioration not attributable to other causes apart from the tumor, per discretion of the treating physician (E) Failure to return for evaluation due to death or deteriorating condition.
Time Frame: 6 months
Population: There were 1 participant in Arm A (cediranib plus olaparib) and 10 participants in Arm B (bevacizumab) that did not receive study treatment. These participants were included in the survival analysis as part of the intention-to-treat population.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Arm A (Olaparib, Cediranib Maleate) | Arm B (Bevacizumab)
Number analyzed (Participants) | 35 | 35
percentage of participants | 16 [5 to 32] | 28 [11 to 47]

2. Secondary Outcome: Progression Free Survival
Description: Progression free survival is defined as the time from randomization until progressive disease or death from any cause.
Time Frame: Up to 3 years
Population: as for outcome 1
Measure: Median (95% Confidence Interval); unit: days
Arm/Group | Arm A (Olaparib, Cediranib Maleate) | Arm B (Bevacizumab)
Number analyzed (Participants) | 35 | 35
days | 118 [63 to 173] | 92 [45 to 142]

3. Secondary Outcome: Overall Survival (OS)
Description: Overall Survival (OS) is defined as the time from randomization to death due to any cause, or censored at date last known alive.
Time Frame: up to 3 years
Population: as for outcome 1
Measure: Median (95% Confidence Interval); unit: days
Arm/Group | Arm A (Olaparib, Cediranib Maleate) | Arm B (Bevacizumab)
Number analyzed (Participants) | 35 | 35
days | 316 [178 to 459] | 218 [135 to 368]

4. Secondary Outcome: Incidence of Adverse Events (AE)
Description: The grade of adverse events be assessed by National Cancer Institute Common Terminology Criteria for Adverse Events 5.0. The incidence of an adverse event at a particular grade is the number of patients who experienced that adverse event/grade.
Time Frame: Up to 3 years
Measure: Count of Participants; unit: Participants
Arm/Group | Arm A (Olaparib, Cediranib Maleate) | Arm B (Bevacizumab)
Number analyzed (Participants) | 34 | 25
Participants
  Anemia: Grade 3 | 2 | 0
  Anemia: Grade 4 | 0 | 0
  Anemia: No grade 3 or above events | 32 | 25
  Leukopenia: Grade 3 | 0 | 0
  Leukopenia: Grade 4 | 1 | 0
  Leukopenia: No grade 3 or above events | 33 | 25
  Neutropenia: Grade 3 | 1 | 0
  Neutropenia: Grade 4 | 1 | 0
  Neutropenia: No grade 3 or above events | 32 | 25
  Lymphopenia: Grade 3 | 2 | 0
  Lymphopenia: Grade 4 | 0 | 0
  Lymphopenia: No grade 3 or above events | 32 | 25
  Thrombocytopenia: Grade 3 | 0 | 1
  Thrombocytopenia: Grade 4 | 1 | 1
  Thrombocytopenia: No grade 3 or above events | 33 | 23
  Hypertension: Grade 3 | 3 | 0
  Hypertension: Grade 4 | 0 | 0
  Hypertension: No grade 3 or above events | 31 | 25
  Heart Failure: Grade 3 | 0 | 0
  Heart Failure: Grade 4 | 1 | 0
  Heart Failure: No grade 3 or above events | 33 | 25
  Transaminitis: Grade 3 | 1 | 0
  Transaminitis: Grade 4 | 0 | 0
  Transaminitis: No grade 3 or above events | 33 | 25
  Intracranial hemorrhage: Grade 3 | 0 | 1
  Intracranial hemorrhage: Grade 4 | 0 | 0
  Intracranial hemorrhage: No grade 3 or above events | 34 | 24
  Muscle weakness of lower limb: Grade 3 | 1 | 0
  Muscle weakness of lower limb: Grade 4 | 0 | 0
  Muscle weakness of lower limb: No grade 3 or above events | 33 | 25
  Hypokalemia: Grade 3 | 2 | 0
  Hypokalemia: Grade 4 | 0 | 0
  Hypokalemia: No grade 3 or above events | 32 | 25
  Thromboembolic event: Grade 3 | 0 | 0
  Thromboembolic event: Grade 4 | 1 | 0
  Thromboembolic event: No grade 3 or above events | 33 | 25
  Dehydration: Grade 3 | 1 | 0
  Dehydration: Grade 4 | 0 | 0
  Dehydration: No grade 3 or above events | 33 | 25
  Paronychia: Grade 3 | 0 | 1
  Paronychia: Grade 4 | 0 | 0
  Paronychia: No grade 3 or above events | 34 | 24

5. Secondary Outcome: Levels of Circulating Cytokines Involved With Angiogenesis
Description: Descriptive statistics will be provided for all continuous biomarkers outcomes. Contingency tables will be provided for categorical data. All comparisons between study arms will be adjusted for multiplicity and in particular false discovery rate (FDR) (Hochberg and Binaymini) will be used for genome data. Binary endpoints will be reported using 95% binomial confidence intervals.
Time Frame: Up to 3 years
Reporting Status: Not Posted, anticipated posting 2025-07

6. Secondary Outcome: Levels of Serial Circulating Biomarkers Involved With Deoxyribonucleic Acid (DNA) Repair
Description: Descriptive statistics will be provided for all continuous biomarkers outcomes. Contingency tables will be provided for categorical data. All comparisons between study arms will be adjusted for multiplicity and in particular FDR (Hochberg and Binaymini) will be used for genome data. Binary endpoints will be reported using 95% binomial confidence intervals.
Time Frame: Up to 3 years
Reporting Status: Not Posted, anticipated posting 2025-07

7. Secondary Outcome: Tumor Genomic Alteration
Description: Will be assessed by whole exome sequencing. Descriptive statistics will be provided for all continuous biomarkers outcomes. Contingency tables will be provided for categorical data. All comparisons between study arms will be adjusted for multiplicity and in particular FDR (Hochberg and Binaymini) will be used for genome data. Binary endpoints will be reported using 95% binomial confidence intervals.
Time Frame: Up to 3 years
Reporting Status: Not Posted, anticipated posting 2025-07

8. Secondary Outcome: Imaging Correlates (Vascular Permeability, Tumor Perfusion and Oxygenation, Brain Tumor Cellularity)
Description: as for outcome 6
Time Frame: Up to 3 years
Reporting Status: Not Posted, anticipated posting 2025-07

ADVERSE EVENTS:
Time Frame: Up to 3 years
Description: All participants who receive at least one dose of cediranib, olaparib or bevacizumab will be evaluable for toxicity from the time of their first treatment. Toxicities will be graded via CTCAE 4.0 until March 31, 2018. CTCAE version 5.0 will be utilized for AE reporting beginning April 1, 2018.
  There were 10 participants in Arm A (cediranib plus olaparib) and 1 participant in Arm B (bevacizumab) that did not receive study treatment, thus were excluded from reporting.
Arm/Group | Arm A (Olaparib, Cediranib Maleate) | Arm B (Bevacizumab)
All-Cause Mortality (participants affected / at risk) | 31/35 | 23/35
Serious Adverse Events (participants affected / at risk) | 16/34 | 13/25
Other Adverse Events (participants affected / at risk) | 33/34 | 24/25
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Arm A (Olaparib, Cediranib Maleate) (N=34) | Arm B (Bevacizumab) (N=25)
Heart Failure (Cardiac disorders) | 1 | 0
Death, not otherwise specified (General disorders) | 1 | 0
Fever (General disorders) | 1 | 0
Esophagitis (Gastrointestinal disorders) | 1 | 0
Neutrophil count decreased (Investigations) | 1 | 0
White blood cell decreased (Investigations) | 1 | 0
Dehydration (Metabolism and nutrition disorders) | 1 | 1
Muscle weakness lower limb (Musculoskeletal and connective tissue disorders) | 1 | 0
Neoplasms - Other - Disease Progression (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2 | 2
Seizure (Nervous system disorders) | 3 | 3
Somnolence (Nervous system disorders) | 1 | 0
Muscle weakness right-sided (Musculoskeletal and connective tissue disorders) | 1 | 0
Muscle weakness left-sided (Musculoskeletal and connective tissue disorders) | 1 | 1
Confusion (Psychiatric disorders) | 1 | 0
Erythema multiforme (Skin and subcutaneous tissue disorders) | 1 | 0
Thromboembolic event (Vascular disorders) | 1 | 0
Cholecystitis (Hepatobiliary disorders) | 0 | 1
Infections & infestations - Other - Upper Respiratory Infection (Infections and infestations) | 0 | 1
Joint infection (Infections and infestations) | 0 | 1
Fall (Injury, poisoning and procedural complications) | 0 | 1
Metabolism and nutrition - Other - Diabetes Insipidus (Metabolism and nutrition disorders) | 0 | 1
Dysphasia (Nervous system disorders) | 0 | 1
Intracranial hemorrhage (Nervous system disorders) | 0 | 1
Syncope (Nervous system disorders) | 0 | 1
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Arm A (Olaparib, Cediranib Maleate) (N=34) | Arm B (Bevacizumab) (N=25)
Abdominal distension (Gastrointestinal disorders) | 1 | 0
Abdominal pain (Gastrointestinal disorders) | 2 | 1
Agitation (Psychiatric disorders) | 1 | 0
Akathisia (Nervous system disorders) | 0 | 1
Alkaline phosphatase increased (Investigations) | 1 | 1
Allergic rhinitis (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Alopecia (Skin and subcutaneous tissue disorders) | 2 | 0
ALT increased (Investigations) | 11 | 3
Amnesia (Nervous system disorders) | 2 | 1
Anemia (Blood and lymphatic system disorders) | 6 | 3
Anorexia (Metabolism and nutrition disorders) | 12 | 0
Anxiety (Psychiatric disorders) | 1 | 1
Arthralgia (Musculoskeletal and connective tissue disorders) | 0 | 3
Arthritis (Musculoskeletal and connective tissue disorders) | 0 | 1
AST increased (Investigations) | 3 | 1
Ataxia (Nervous system disorders) | 1 | 0
Back pain (Musculoskeletal and connective tissue disorders) | 0 | 1
Blood bilirubin increased (Investigations) | 3 | 1
Blood/Lymph - Other - Decreased Rbc (Blood and lymphatic system disorders) | 1 | 0
Blood/Lymph - Other - Elevated White Blood Count (Blood and lymphatic system disorders) | 1 | 1
Blood/Lymph - Other - Hyperphosphatemia (Blood and lymphatic system disorders) | 0 | 1
Blood/Lymph - Other - Lft Abnormailities (Blood and lymphatic system disorders) | 0 | 1
Blurred vision (Eye disorders) | 2 | 0
Bruising (Injury, poisoning and procedural complications) | 1 | 0
Cognitive disturbance (Nervous system disorders) | 1 | 2
Concentration impairment (Nervous system disorders) | 1 | 0
Confusion (Psychiatric disorders) | 4 | 3
Constipation (Gastrointestinal disorders) | 4 | 3
Cough (Respiratory, thoracic and mediastinal disorders) | 2 | 4
Creatinine increased (Investigations) | 2 | 0
Dehydration (Metabolism and nutrition disorders) | 1 | 0
Depression (Psychiatric disorders) | 1 | 1
Diarrhea (Gastrointestinal disorders) | 19 | 4
Dizziness (Nervous system disorders) | 6 | 3
Dry eye (Eye disorders) | 2 | 0
Dry mouth (Gastrointestinal disorders) | 1 | 0
Dry skin (Skin and subcutaneous tissue disorders) | 1 | 0
Dysarthria (Nervous system disorders) | 2 | 0
Dysgeusia (Nervous system disorders) | 2 | 0
Dyspepsia (Gastrointestinal disorders) | 4 | 0
Dysphagia (Gastrointestinal disorders) | 3 | 0
Dysphasia (Nervous system disorders) | 3 | 3
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 2 | 0
Ear and Labyrinth - Other - Ears Feeled Stuffed Up Like A Head Cold (Ear and labyrinth disorders) | 1 | 0
Ear pain (Ear and labyrinth disorders) | 2 | 0
Edema face (General disorders) | 1 | 0
Edema limbs (General disorders) | 3 | 0
Edema trunk (General disorders) | 1 | 0
Encephalopathy (Nervous system disorders) | 0 | 1
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Eye disorders - Other, specify - Diplopia (Eye disorders) | 1 | 0
Eye disorders - Other, specify - Left Homonymous Hemianopsia (Eye disorders) | 1 | 0
Eye disorders - Other, specify - Left Sided Field Cut (Eye disorders) | 1 | 0
Facial nerve disorder (Nervous system disorders) | 0 | 1
Fall (Injury, poisoning and procedural complications) | 7 | 5
Fatigue (General disorders) | 12 | 8
Fecal incontinence (Gastrointestinal disorders) | 0 | 2
Fever (General disorders) | 0 | 1
Flank pain (Musculoskeletal and connective tissue disorders) | 1 | 0
Flu like symptoms (General disorders) | 0 | 1
Gait disturbance (General disorders) | 9 | 1
Gastroesophageal reflux disease (Gastrointestinal disorders) | 2 | 1
General and admin site - Other - Abdominal Discomfort (General disorders) | 1 | 0
General and admin site - Other - Decreased Dexterity (General disorders) | 1 | 0
General and admin site - Other - Double Vision (General disorders) | 1 | 0
General and admin site - Other - Executive Dysfunction (General disorders) | 1 | 0
General and admin site - Other - Failure To Thrive (General disorders) | 1 | 0
General and admin site - Other - Mood Swings (General disorders) | 1 | 0
General and admin site - Other - Ptosis (General disorders) | 1 | 0
General and admin site - Other - Temperature Intolerance (General disorders) | 1 | 0
General and admin site - Other - Voice Hoarseness (General disorders) | 1 | 0
Generalized muscle weakness (Musculoskeletal and connective tissue disorders) | 2 | 3
GI disorders - Other, specify - Belching (Gastrointestinal disorders) | 1 | 0
GI disorders - Other, specify - Dysuria (Gastrointestinal disorders) | 1 | 0
GI disorders - Other, specify - Gi Virus (Gastrointestinal disorders) | 1 | 0
Headache (Nervous system disorders) | 8 | 4
Hematuria (Renal and urinary disorders) | 2 | 4
Hemorrhoidal hemorrhage (Gastrointestinal disorders) | 1 | 0
Hiccups (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Hoarseness (Respiratory, thoracic and mediastinal disorders) | 2 | 3
Hypercalcemia (Metabolism and nutrition disorders) | 0 | 1
Hyperglycemia (Metabolism and nutrition disorders) | 2 | 3
Hyperhidrosis (Skin and subcutaneous tissue disorders) | 1 | 0
Hyperkalemia (Metabolism and nutrition disorders) | 3 | 2
Hypersomnia (Nervous system disorders) | 2 | 0
Hypertension (Vascular disorders) | 21 | 7
Hyperthyroidism (Endocrine disorders) | 0 | 2
Hyperthyroidism (Metabolism and nutrition disorders) | 1 | 0
Hypocalcemia (Metabolism and nutrition disorders) | 0 | 2
Hypoglycemia (Metabolism and nutrition disorders) | 1 | 1
Hypokalemia (Metabolism and nutrition disorders) | 4 | 1
Hyponatremia (Metabolism and nutrition disorders) | 5 | 2
Hypophosphatemia (Metabolism and nutrition disorders) | 2 | 1
Hypotension (Vascular disorders) | 1 | 1
Hypothyroidism (Endocrine disorders) | 7 | 2
Infections & infestations - Other - Flu Symptoms (Infections and infestations) | 0 | 1
Infections & infestations - Other - Muscal (Infections and infestations) | 1 | 0
Infections & infestations - Other - Thrush (Infections and infestations) | 3 | 0
Infections & infestations - Other - Upper Respiratory Infection (Infections and infestations) | 0 | 1
Injury/poison/procedure - Other - Ear Laceration (Injury, poisoning and procedural complications) | 0 | 1
Insomnia (Psychiatric disorders) | 2 | 1
Intracranial hemorrhage (Nervous system disorders) | 1 | 1
Investigations - Other, specify - Cerebral Edema (Investigations) | 0 | 1
Irritability (Psychiatric disorders) | 0 | 1
Joint range of motion decreased (Musculoskeletal and connective tissue disorders) | 0 | 1
Lethargy (Nervous system disorders) | 0 | 1
Localized edema (General disorders) | 0 | 1
Lymphocyte count decreased (Investigations) | 5 | 4
Memory impairment (Nervous system disorders) | 3 | 1
Metabolism and nutrition - Other - Diabetes Insipidus (Metabolism and nutrition disorders) | 0 | 1
Metabolism and nutrition - Other - Liver Function Tests Elevated (Metabolism and nutrition disorders) | 1 | 0
Mucosal infection (Infections and infestations) | 1 | 0
Mucositis oral (Gastrointestinal disorders) | 4 | 0
Muscle weakness left-sided (Nervous system disorders) | 4 | 4
Muscle weakness lower limb (Musculoskeletal and connective tissue disorders) | 3 | 3
Muscle weakness right-sided (Nervous system disorders) | 0 | 1
Musculoskel/connect tissue -Other - Muscle Cramp (Musculoskeletal and connective tissue disorders) | 1 | 0
Myalgia (Musculoskeletal and connective tissue disorders) | 0 | 2
Nasal congestion (Respiratory, thoracic and mediastinal disorders) | 0 | 2
Nausea (Gastrointestinal disorders) | 12 | 1
Neoplasms - Other - Disease Progression (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Neoplasms - Other - Labial Cyst (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Neoplasms - Other - Tubular Adenoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Nervous system - Other - Aphasia (Nervous system disorders) | 1 | 0
Nervous system - Other - Left 6th Palsy (Nervous system disorders) | 1 | 0
Nervous system - Other - Left Eye Ptosis (Nervous system disorders) | 1 | 0
Nervous system - Other - Right Tongue Deviation (Nervous system disorders) | 1 | 0
Neutrophil count decreased (Investigations) | 5 | 1
Non-cardiac chest pain (General disorders) | 1 | 0
Oral dysesthesia (Gastrointestinal disorders) | 1 | 0
Pain (General disorders) | 3 | 2
Pain in extremity (Musculoskeletal and connective tissue disorders) | 1 | 2
Paresthesia (Nervous system disorders) | 2 | 1
Paronychia (Infections and infestations) | 0 | 1
Peripheral motor neuropathy (Nervous system disorders) | 1 | 0
Personality change (Psychiatric disorders) | 1 | 1
Platelet count decreased (Investigations) | 10 | 8
Postnasal drip (Respiratory, thoracic and mediastinal disorders) | 2 | 0
PPE syndrome (Skin and subcutaneous tissue disorders) | 2 | 0
Premature menopause (Reproductive system and breast disorders) | 0 | 1
Proteinuria (Renal and urinary disorders) | 7 | 7
Pyramidal tract syndrome (Nervous system disorders) | 1 | 0
Rash acneiform (Skin and subcutaneous tissue disorders) | 1 | 1
Rash maculo-papular (Skin and subcutaneous tissue disorders) | 1 | 0
Resp, thoracic & mediast - Other - Tan Phlegm (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Seizure (Nervous system disorders) | 6 | 1
Sinus bradycardia (Cardiac disorders) | 1 | 1
Sinus pain (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Sinus tachycardia (Cardiac disorders) | 1 | 1
Sinusitis (Infections and infestations) | 1 | 0
Skin & subcutaneous tissue -Other - Abrasion (Skin and subcutaneous tissue disorders) | 1 | 0
Skin & subcutaneous tissue -Other - Lesion, L Upper Arm, L Groin (Skin and subcutaneous tissue disorders) | 0 | 1
Skin & subcutaneous tissue -Other - Rash, Nos (Skin and subcutaneous tissue disorders) | 0 | 1
Skin infection (Infections and infestations) | 1 | 1
Skin infection (Skin and subcutaneous tissue disorders) | 0 | 1
Somnolence (Nervous system disorders) | 1 | 0
Sore throat (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Stomach pain (Gastrointestinal disorders) | 1 | 0
Surgical and medical - Other - L True Voal Cord Medialization With Prolaryn Hydroxyapalite (Surgical and medical procedures) | 0 | 1
Surgical and medical - Other - Left True Vocal Cord Medialization With Prolaryn Hydroxyapatite (Surgical and medical procedures) | 0 | 1
Surgical and medical - Other - Lumbar Radiculopathy (Surgical and medical procedures) | 0 | 2
Thromboembolic event (Vascular disorders) | 1 | 0
Tooth infection (Infections and infestations) | 0 | 1
Toothache (Gastrointestinal disorders) | 1 | 1
Tremor (Nervous system disorders) | 2 | 0
Upper respiratory infection (Infections and infestations) | 2 | 2
Urinary incontinence (Renal and urinary disorders) | 1 | 0
Urinary tract infection (Infections and infestations) | 31 | 1
Urinary urgency (Renal and urinary disorders) | 1 | 0
Vertigo (Ear and labyrinth disorders) | 1 | 0
Vomiting (Gastrointestinal disorders) | 8 | 0
Weight gain (Investigations) | 0 | 2
Weight loss (Investigations) | 6 | 0
White blood cell decreased (Investigations) | 5 | 4
Wound dehiscence (Injury, poisoning and procedural complications) | 0 | 1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of 60 days or less

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2019-05-10): https://cdn.clinicaltrials.gov/large-docs/21/NCT02974621/Prot_SAP_000.pdf